CLINICAL TRIAL: NCT04220788
Title: Pharmacist Enhanced Service in Primary Care for CArdiovascular Risk Reduction (PxES-CAR2+) Project: A Multi-centre Pragmatic, Step-wedge Cluster Randomized Controlled Trial
Brief Title: Pharmacist Enhanced Service for Cardiovascular Risk Reduction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment due to difficulty in recruitment of study sites
Sponsor: Monash University (Other)
Collaborators: Klinik Kesihatan Puchong (Unknown); Klinik Kesihatan Kelana Jaya (Unknown); Klinik Kesihatan Shah Alam Seksyen 7 (Unknown); Klinik Kesihatan Shah Alam Seksyen 9 (Unknown); Klinik Kesihatan Taman Medan (Unknown); Klinik Kesihatan Seri Kembangan (Unknown)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Associate Professor, Monash University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: PxES-CAR2+
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Risk Factor
Keywords: cardiovascular disease; pharmacist service
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced pharmacist service (Experimental): The advanced care group will be undergo a Comprehensive Annual Care Plan (CACP) or Standard Medication Management Assessment (SMMA) with the pharmacist
  Interventions: Other: Enhanced pharmacist service
- Usual care (Active Comparator): Patients in the usual care arm will receive their usual care which they will obtain care from their doctor,nurse and pharmacist where appropriate
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Enhanced pharmacist service — Calculation of cardiovascular risk by an online tool for discussion on the CVD risk. Pharmacist will also provide ducation on cardiovascular risk factors and healthy lifestyle. Any prescription adaptation(s), and/or recommendations where necessary to meet lipid, blood pressure and glycemic control targets and smoking cessation will be initiated
  Arms: Enhanced pharmacist service
Other: Usual care — Participants in the arm will receive their care from their respective nurse, doctor or pharmacists as per usual clinic practice
  Arms: Usual care

SUMMARY:
Pharmacist services such as medication review, counselling and treatment adherence clinics can improve clinical, health related quality of life and economic outcomes. To prove this hypothesis a step-wedge, cluster randomized controlled trial will be held in primary care centers of the public health system of Malaysia. Participants who have a high risk of cardiovascular risk factors currently seeking care in primary care will be recruited. Control group will receive usual care and the intervention arm will be seen by a pharmacist prior to their follow-up, with a comprehensive medication review, counselling and dietary advice consultations every month for three months. Participating pharmacist will be trained in cardiovascular prevention pharmacotherapy, interview skills, educational techniques, and develop personalized plan for every participant. The investigators plan to randomize up to 2100 participants who are currently receiving care in the primary care clinics in the district of Petaling by modifying the current workflow in primary care, whereby the investigators aim to get participants who are at high risk to undergo counselling as well as a medication review with proper pharmaceutical care delivered to them prior to seeking their medical doctor to receive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes
* Patients with chronic kidney disease (eGFR <60ml/min/1.73m2)
* Patients with established atherosclerotic vascular disease (via patient health records or selfreport) including cerebrovascular disease (prior stroke or transient ischemic attack), cardiovascular disease (myocardial infarction, acute coronary syndrome, stable angina, or revascularization), or peripheral arterial disease (symptomatic and/or ankle brachial index <0.9)
* Primary prevention patients with multiple risk factors and Framingham risk score >30%

Exclusion Criteria:

* Unwilling to participate/sign consent form
* Unwilling or unable to participate in regular follow-up visits
* Pregnancy
* Undergoing existing medication therapy adherence clinic conducted by the Pharmacy Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cardiovascular risk scores | 3 months
  The difference from baseline to 3 months in the estimated cardiovascular risk between advanced care and usual care groups assessed using the Framingham scale

SECONDARY OUTCOMES:
Change in cardiovascular risk scores | 6 months
  The difference from baseline to 6 months in the estimated cardiovascular risk between advanced care and usual care groups assessed using the Framingham scale
Change in cardiovascular risk scores | 12 months
  The difference from baseline to 12 months in the estimated cardiovascular risk between advanced care and usual care groups assessed using the Framingham scale
Change in cardiovascular risk scores | 24 months
  The difference from baseline to 24 months in the estimated cardiovascular risk between advanced care and usual care groups assessed using the Framingham scale
Achievement of recommended cholesterol, blood pressure and glycemic control targets | 3 months
  Number of individual achieving target cholesterol, blood pressure and glycemic control target
Proportion of patients receiving appropriate medication | 3 months
  Number of patients receiving appropriate BP, cholesterol and diabetes medication

OTHER OUTCOMES:
Efficiency of screening | 3 months
  Number of high risk patients screened for cardiovascular risk
Change in participant quality of life | 3 months
  Change in quality of life assessed using EuroQoL-5D from baseline to end of intervention (range 0-1)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Lee, Principal Investigator — Monash University Malaysia
Locations (1):
- Shaun Lee, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No